CLINICAL TRIAL: NCT00137540
Title: First Line Radiofrequency Ablation vs. Antiarrhythmic Drugs for Atrial Fibrillation Treatment
Brief Title: FLAT Study: First Line Ablation Therapy for Treatment of Paroxysmal Atrial Fibrillation (RAAFT)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biosense Webster EMEA (Industry)
Responsible Party: Sponsor
Organization: Biosense Webster, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FLAT
Record Dates: First submitted 2005-08-29; First posted 2005-08-30 (Estimated); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Atrial Fibrillation
Keywords: First line ablation therapy
MeSH Terms: conditions — Atrial Fibrillation

INTERVENTIONS:
Device: RF ablation
Drug: anti-arrhythmic drug therapy

SUMMARY:
The objective of this multicenter randomized study is to establish the effectiveness of treatment for paroxysmal atrial fibrillation (AF), in patients not previously treated with anti-arrhythmic drugs, by encircling the pulmonary veins with radiofrequency (RF) ablation, using the NaviStar® ThermoCool® catheter and the CARTO™ EP Navigation System. Effectiveness will be determined by comparing chronic success of ablation therapy versus anti-arrhythmic drug treatment, defined as patients with an absence of atrial tachycardias during 24 months of follow-up as determined by 7-days Holter and transtelephonic monitoring, and by 12-lead electrocardiogram (ECG) recordings.

DETAILED DESCRIPTION:
This study is a prospective, randomized, multicenter clinical study that will enroll in its first phase 40 patients. The study will be performed in 3 European hospitals. Patients will be randomized to either the RF ablation strategy or to the medication arm.

Hypothesis:

As first line therapy, catheter ablation improves the long-term success, health-economic outcomes and is equally safe compared to the best anti-arrhythmic medication treatment in a selected group of patients with paroxysmal atrial fibrillation.

Primary endpoint:

* long-term success, defined as patients free from any atrial fibrillation during 24 months after initial study treatment as determined by 7-days Holter and transtelephonic monitoring and by 12-lead ECG recordings.

Secondary endpoints:

* AF burden: frequency and duration of episodes
* health-economic costs over 24 months
* serious adverse events
* Quality of Life scores, using SF-36 questionnaire

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained
* Two or more documented symptomatic paroxysmal atrial fibrillation episodes during the last 6 months. Episodes should last longer than 30 seconds.
* Patients should not be on anti-arrhythmic medication therapy (Class I, III or IV) for AF (other than for cardioversion) or are currently on antiarrhythmic drug (AAD) therapy for any other arrhythmia

Exclusion Criteria:

* Patients who had a previous ablation for atrial fibrillation
* Patients who had presence of severe valvular disease, myocardial infarction and/ or cardiomyopathy
* Patients with a left atrial size more than 50 mm
* Patients who had more than 2 cardioversions
* Patients who have a history of AF for less than 3 months or more than one year
* Patients with solely asymptomatic AF
* Patients who have AF episodes triggered by another uniform arrhythmia
* Patients who actively abuse alcohol or other drugs, which may be causative of AF
* Patients with a tumor, or another abnormality which precludes catheter introduction
* Patients with a revascularization or other cardiac surgery within 6 months before study treatment
* Patients in whom appropriate vascular access is precluded
* Patients with a contraindication to treatment with warfarin or other bleeding diathesis participants in another investigational clinical or device trial
* Patients who are inaccessible for follow-up psychological problem that might limit compliance
* Patients who cannot or will not fulfill the follow-up or protocol requirements
* Pregnant women
* Patients with severe chronic obstructive pulmonary disease
* Patients with Wolff-Parkinson-White (WPW) syndrome
* Patients with renal failure requiring dialysis
* Patients with hepatic failure

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2005-09; Primary Completion 2007-04 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
long-term success | 19 months

SECONDARY OUTCOMES:
AF-burden | 19 months
health-economic costs | 24 months
serious adverse events | 19 months
Quality of Life scores | 19 months

CONTACTS AND LOCATIONS:
Overall Officials: F. Gaita, Prof., Principal Investigator — Ospedale Civile, Asti, Italy; P. Della Bella, MD, Principal Investigator — Centro Cardiologico Monzino, Milan, Italy; M. Fiala, MD, Principal Investigator — Nemocnice Podlesi, Trinec, Czech Republic